CLINICAL TRIAL: NCT00227136
Title: Effect of Oral 5-HTP Intake on Urinary 5-HIAA Excretion
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Organization: Western University, Canada (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 5-HTPSVU
Record Dates: First submitted 2005-09-23; First posted 2005-09-27 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2006-07

CONDITIONS: Carcinoid Tumors; Neuroendocrine Tumors
Keywords: 5Hydroxytryptamine; Chromogranin A; 5HIAA; carcinoid
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors | interventions — Serotonin

INTERVENTIONS:
Drug: 5-Hydroxy-Tryptamine

SUMMARY:
This is a research study looking at the effect of 5-Hydroxy Tryptophan (5-HTP) on urine excretion of 5-Hydroxyindolacetic acid (5-HIAA). 5-HTP is a common over the counter product that is sold in natural food stores and via the Internet. Increased levels of 5-HIAA in the urine can be found in a specific type of cancer, called carcinoid tumor. This study will examine the effect of oral 5-HTP intake on 5-HIAA excretion. Understanding this effect may help to determine which tests should be done in a patient with increased 5-HIAA excretion who's also taking 5-HTP.

DETAILED DESCRIPTION:
5-HTP is a common over the counter product that is sold in natural food stores and via the Internet. It is claimed to improve sleep problems, depression, anxiety, compulsive disorders, restless leg syndrome, migraines, fibromyalgia, and low pain threshold.Increased levels of 5-HIAA in the urine can be a of a specific type of cancer, called carcinoid tumor. Urinary 5-HIAA levels can also be increased by a number of food products and drugs. Oral 5-HTP is not known as a cause of elevation of 5-HIAA in urine. However, recent information suggests that 5-HTP may cause an increase.

In this study we examine the effect of oral 5-HTP intake (100 mg at bedtime for 10 days) on 5-HIAA excretion in the urine, following a prospective, double-blind placebo-controlled study design.

Understanding this effect may help to determine which tests should be done in a patient with increased 5-HIAA excretion who's also taking 5-HTP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* in good health

Exclusion Criteria:

* Pregnancy
* Intake of drugs that affect 5-HIAA excretion in urine
* Anti-depressants
* Participation in other studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2005-05; Study Completion 2005-09

PRIMARY OUTCOMES:
Urinary excretion of 5-HIAA
Plasma Chromogranin A

SECONDARY OUTCOMES:
Side effects

CONTACTS AND LOCATIONS:
Overall Officials: Stan HM Van Uum, MD, PhD, Principal Investigator — Western University, Canada
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada